CLINICAL TRIAL: NCT07330102
Title: Systematic Approach for Cold Knife Morcellation of Large Uterus in Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 368
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Hysterectomy, Benign Uterine Diseases
Keywords: Hysterectomy; Morcellation; Large uterus
MeSH Terms: interventions — Morcellation

STUDY DESIGN:
Intervention Model Description: Following the completion of the TLH and before vault closure, the uterus is flipped upside down to resemble a flask and is grasped by the assistant from the cervix. The endoknife is advanced carefully through a 10 mm trocar and an incision is started from the level of the isthmus and advanced sagittally towards the fundus to bisect this uterus into two hemiuteri connected at the fundus. The incision is stopped 1-2 cm before the fundus to keep the specimen intact. The uterus (which is grasped from the cervix) is then rotated 90 degrees and another incision is started in the hemiuterus containing the cervix coronally towards the fundus again bisecting this hemiuterus. The incision is advanced through the connecting fundus bisecting the other hemiuterus. The incision is stopped 1-2 cm before the specimen is split into two. The end result is a long, connected strip of uterus formed of the bisected hemiuteri.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morecellation group (Experimental): Morcellation of the large uterus
  Interventions: Procedure: Morcellation

INTERVENTIONS:
Procedure: Morcellation — Following the completion of the TLH and before vault closure, the uterus is flipped upside down to resemble a flask and is grasped by the assistant from the cervix. The endoknife is advanced carefully through a 10 mm trocar and an incision is started from the level of the isthmus and advanced sagittally towards the fundus to bisect this uterus into two hemiuteri connected at the fundus. The incision is stopped 1-2 cm before the fundus to keep the specimen intact. The uterus (which is grasped from the cervix) is then rotated 90 degrees and another incision is started in the hemiuterus containing the cervix coronally towards the fundus again bisecting this hemiuterus. The incision is advanced through the connecting fundus bisecting the other hemiuterus. The incision is stopped 1-2 cm before the specimen is split into two. The end result is a long, connected strip of uterus formed of the bisected hemiuteri.

SUMMARY:
Following the completion of the TLH and before vault closure, the uterus is flipped upside down to resemble a flask and is grasped by the assistant from the cervix. The endoknife is advanced carefully through a 10 mm trocar and an incision is started from the level of the isthmus and advanced sagittally towards the fundus to bisect this uterus into two hemiuteri connected at the fundus. The incision is stopped 1-2 cm before the fundus to keep the specimen intact. The uterus (which is grasped from the cervix) is then rotated 90 degrees and another incision is started in the hemiuterus containing the cervix coronally towards the fundus again bisecting this hemiuterus. The incision is advanced through the connecting fundus bisecting the other hemiuterus. The incision is stopped 1-2 cm before the specimen is split into two. The end result is a long, connected strip of uterus formed of the bisected hemiuteri. The cervix is guided through the colpotomy and is grasped vaginally with a tenaculum and pulled exteriorly. The vault is then closed with a continuous suture.

DETAILED DESCRIPTION:
Following the completion of the TLH and before vault closure, the uterus is flipped upside down to resemble a flask and is grasped by the assistant from the cervix. The endoknife is advanced carefully through a 10 mm trocar and an incision is started from the level of the isthmus and advanced sagittally towards the fundus to bisect this uterus into two hemiuteri connected at the fundus. The incision is stopped 1-2 cm before the fundus to keep the specimen intact. The uterus (which is grasped from the cervix) is then rotated 90 degrees and another incision is started in the hemiuterus containing the cervix coronally towards the fundus again bisecting this hemiuterus. The incision is advanced through the connecting fundus bisecting the other hemiuterus. The incision is stopped 1-2 cm before the specimen is split into two. The end result is a long, connected strip of uterus formed of the bisected hemiuteri. The cervix is guided through the colpotomy and is grasped vaginally with a tenaculum and pulled exteriorly. The vault is then closed with a continuous suture.

ELIGIBILITY:
Inclusion Criteria:

* Women candidates for total laparoscopic hysterectomy
* Uterus size >/= 20 weeks gravid uterus
* Benign uterine disease

Exclusion Criteria:

* • Malignant or premalignant uterine disease
* Bleeding disorders
* Unfit for surgery
* Contraindications for laparoscopy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Time of operation | At time of surgery
  Total time of the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided